CLINICAL TRIAL: NCT04996017
Title: PHASE III STUDY WITH ATEZOLIZUMAB VERSUS PLACEBO IN MALIGNANT PLEURAL MESOTHELIOMA PATIENTS AFTER PLEURECTOMY/DECORTICATION
Brief Title: Atezolizumab Versus Placebo for the Adjuvant Treatment of Malignant Pleural Mesothelioma (Atezomeso)
Acronym: AtezoMeso
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Gruppo Oncologico Italiano di Ricerca Clinica (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GOIRC -03-2019
Record Dates: First submitted 2021-05-25; First posted 2021-08-09 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Mesotheliomas Pleural
Keywords: mesothelioma; Adjuvant therapy; immunotherapy
MeSH Terms: conditions — Mesothelioma, Malignant; Mesothelioma | interventions — atezolizumab; Injections

STUDY DESIGN:
Intervention Model Description: This is a multicentric double-blind, placebo controlled, phase III trial. In this study, patients who underwent to a surgical resection of pleural mesothelioma and are without signs of macroscopic residual disease will be randomized 2:1 to receive atezolizumab or placebo. Patients will be treated for 12 months or until recurrence, unacceptable toxicity or patient/physician decision, whichever occurs first. Randomization will be done via a centralized system and patients will be stratified histology (epithelioid vs non epithelioid) and stage (I vs
  >I).
Who Masked: Care Provider
Masking Description: This is a randomized, placebo-controlled, double-blind study. Patients will be randomized to one of the following treatment arms in a 2:1 ratio (experimental to control arm):
  * Arm A (experimental arm): atezolizumab
  * Arm B (control arm): placebo
  Randomization will be stratified by the following factors:
  * Histology (epithelioid vs non epithelioid)
  * Stage (I vs >I) Blinding Investigators and patients will remain blinded to treatment assignment until the final analysis of OS, except in the event unblinding is necessary for a medical emergency or to help guide decisions on subsequent treatment.
  If the investigator wishes to know the identity of the study drug for any reason other than a medical emergency, he or she should contact the Scientific Responsible. In case of unblinding, patient will be withdrawn by the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): atezolizumab 1200mg every 21 days
  Interventions: Drug: Atezolizumab 1200 mg in 20 ML Injection
- Arm B (Placebo Comparator): Placebo will be supplied by the sponsor and will be identical in appearance to atezolizumab and will comprise the same excipients but without atezolizumab every 21 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Atezolizumab 1200 mg in 20 ML Injection — Atezolizumab will be supplied as sterile liquid in 20-mL glass vials. The vial is designed to deliver 20 mL (1200 mg) of atezolizumab solution but may contain more than the stated volume to enable delivery of the entire 20 mL volume. For information on the formulation and handling of atezolizumab, refer to the Atezolizumab Investigator's Brochure.
  Arms: Arm A
Drug: Placebo — Placebo will be supplied as sterile liquid in 20ml vials. the vial is designed
  Arms: Arm B

SUMMARY:
This is a multicentric double-blind, placebo controlled, phase III trial. In this study, patients who underwent to a surgical resection of pleural mesothelioma and are without signs of macroscopic residual disease will be randomized 2:1 to receive atezolizumab or placebo. Patients will be treated for 12 months or until recurrence, unacceptable toxicity or patient/physician decision, whichever occurs first.

Randomization will be done via a centralized system and patients will be stratified histology (epithelioid vs non epithelioid) and stage (I vs

>I). Patients will be radiologically evaluated after surgical procedure before starting therapy and then every 12 weeks for 24 months or until disease progression. At screening patients should be without macroscopic residual disease. Quality of life questionnaire will be administered to patient at baseline and every 12 weeks. During the study baseline tumor blocks will be centrally analyzed to determinate biological characteristics and gene expression.

ELIGIBILITY:
Inclusion Criteria

* Signed informed Consent Form
* Age ≥ 18 years on day of signing informed consent
* Histologically confirmed malignant pleural mesothelioma
* Surgical resection (P/D), without macroscopic residual. For stage I patient without visceral involvement a total pleurectomy is allowed
* Absence of measurable or non-measurable disease assessed with CT scan after surgery
* Patients must have received at least no 4 cycles of platinum/pemetrexed
* perioperative chemotherapy as per local practice (neoadjuvant or adjuvant or both). Less than 4 cycles of chemotherapy are allowed for clinical decisions

  - In patients previously treated with neoadjuvant chemotherapy, randomization
* should occur within 50 days from surgical resection.

  - In patients treated with adjuvant chemotherapy, randomization should occur
* within 30 ±7 days from last dose of adjuvant treatment.
* Performance status of 0-1 on the ECOG Performance Scale
* Availability of a representative tumor specimen for exploratory biomarker research (see Section 4.5.6 for information on tumor specimens) A formalin-fixed paraffin-embedded (FFPE) tumor specimen in a paraffin block (preferred) or at least 10 slides containing unstained, freshly cut, serial sections must be submitted along with an associated pathology report prior to study enrollment.
* Adequate hematologic and end-organ function, defined by the following laboratory test results, obtained within 14 days prior to initiation of study treatment: ANC ³ 1.5 ´ 109/L (1500/mL) without granulocyte colony-stimulating factor support Lymphocyte count ³ 0.5 ´ 109/L (500/mL) Platelet count ³ 100 ´ 109/L (100,000/mL) without transfusion Hemoglobin 9 g/dL Patients may be transfused to meet this criterion. AST, ALT, and alkaline phosphatase (ALP) £ 2.5 ´ upper limit of normal (ULN)

Bilirubin £ 1.5 ´ ULN with the following exception:

Patients with known Gilbert disease: bilirubin level £ 3 ´ ULN. Creatinine £ 1.5 ´ ULN Albumin ³ 25 g/L (2.5 g/dL) For patients not receiving therapeutic anticoagulation: INR or aPTT £ 1.5 ´ ULN

• For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraception, as defined below: Women must remain abstinent or use contraceptive methods with a failure rate of < 1% per year during the treatment period and for 5 months after the final dose of atezolizumab. Women must refrain from donating eggs during this same period.

A woman is considered to be of childbearing potential if she is postmenarcheal, hasnot reached a postmenopausal state (³12 continuous months of amenorrhea with no identified cause other than menopause), and is not permanently infertile due to surgery (i.e., removal of ovaries, fallopian tubes, and/or uterus) or another cause as determined by the investigator (e.g., Müllerian agenesis). Examples of contraceptive methods with a failure rate of <1% per year include bilateral tubal ligation, male sterilization, hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices.

The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) andn withdrawal are not acceptable methods of contraception. If required per local guidelines or regulations, locally recognized acceptable methods of contraception and information about the reliability of abstinence will be described in the local Informed Consent Form.

Women with a positive pregnancy test at enrollment or prior to administration of study medication will be excluded.

Exclusion Criteria

* Patient with macroscopic residual disease after surgery, evaluated with CT scan
* after surgery or adjuvant therapy
* Subjects with active, known or suspected autoimmune disease. Subjects with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll
* Additional malignancy in the last 5 years. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy
* Active infection requiring systemic therapy
* Patient with positive result to Human Immunodeficiency Virus (HIV) (HIV 1/2
* antibodies) test
* Active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected) 7. History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis
* obliterans), drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of
* active pneumonitis on screening chest computed tomography (CT) scan. NOTE:
* History of radiation pneumonitis in the radiation field (fibrosis) is permitted
* Known active tuberculosis
* Significant cardiovascular disease (such as New York Heart Association Class II or
* greater cardiac disease, myocardial infarction, or cerebrovascular accident) within 3 months prior to initiation of study treatment, unstable arrhythmia, or unstable
* angina
* Major surgical procedure, other than for diagnosis, within 4 weeks prior to initiation of
* study treatment, or anticipation of need for a major surgical procedure during the
* study
* Severe infection within 4 weeks prior to initiation of study treatment, including, but
* not limited to, hospitalization for complications of infection, bacteremia, or severe
* pneumonia
* Prior allogeneic stem cell or solid organ transplantation
* Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that contraindicates the use of an investigational drug, may affect the interpretation of the results, or may render the patient at high risk from treatment complications
* Treatment with a live, attenuated vaccine within 4 weeks prior to initiation of study treatment, or anticipation of need for such a vaccine during atezolizumab treatment or within 5 months after the final dose of atezolizumab15. Current treatment with anti-viral therapy for HBV
* Treatment with investigational therapy within 28 days prior to initiation of study
* treatment
* Prior treatment with CD137 agonists or immune checkpoint blockade therapies, including anti-CTLA-4, anti-PD-1, and anti-PD-L1 therapeutic antibodies
* Treatment with systemic immunostimulatory agents (including, but not limited to, interferon and interleukin 2 [IL-2]) within 4 weeks or 5 drug elimination half-lives (whichever is longer) prior to initiation of study treatment
* Treatment with systemic immunosuppressive medication (including, but not limited to, corticosteroids, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-TNF-a agents) within 2 weeks prior to initiation of study treatment, or anticipation of need for systemic immunosuppressive medication during study treatment, with the following exceptions:

  * Patients who received acute, low-dose systemic immunosuppressant medication or a one-time pulse dose of systemic immunosuppressant medication (e.g., 48 hours of corticosteroids for a contrast allergy) are eligible for the study after Scientific Responsible approval has been obtained
  * Patients who received mineralocorticoids (e.g., fludrocortisone), corticosteroids for chronic obstructive pulmonary disease (COPD) or asthma, or low-dose corticosteroids for orthostatic hypotension or adrenal insufficiency are eligible for the study
* History of severe allergic anaphylactic reactions to chimeric or humanized antibodies or fusion proteins
* Known hypersensitivity to Chinese hamster ovary cell products or to any component of the atezolizumab formulation
* Pregnancy or breastfeeding, or intention of becoming pregnant during study treatment or within 5 months after the final dose of study treatment
* Women of childbearing potential must have a negative serum pregnancy test result within 14 days prior to initiation of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2021-12-14 (Actual); Primary Completion 2027-07-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
To evaluate the efficacy of atezolizumab in patients with MPM in terms of DFS | 12 weeks
  DFS, defined as the time from initiation of study treatment to first recurrence of disease or death for any cause, whichever occurs first.

SECONDARY OUTCOMES:
To evaluate the safety of atezolizumab in patients with MPM | 12 months
  Incidence, nature, frequency, duration, timing and severity of serious adverse events (SAEs) and non-serious adverse events (AEs) related to atezolizumab treatment graded by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v. 5.
To evaluate the efficacy of atezolizumab in patients with MPM in terms of OS | 12 months
  OS, defined as the time from start of study drug to the date of death from any cause

CONTACTS AND LOCATIONS:
Locations (19):
- Italy (19):
  - Istituto Scientifico Romagnolo Per Lo Studio E La Cura Dei Tumori - Irccs, Meldola, ITAòY
  - Ospedaliera SS Antonio e Biagio e Cesare Arrigo di Alessandria, Alessandria
  - Istituto Tumori Bari, Bari
  - Azienda Ospedaliera Universitaria Policlinico- Vittorio Emanuele Catania, Catania
  - Ospedale Ss Annunziata, Chieti
  - Azienda Ospedaliero Universitaria di Ferrara, Ferrara
  - Villa Scassi, Genova
  - Ospedale Dell'Angelo, Mestre
  - Azienda Ospedaliera Universitaria Di Modena, Modena
  - Aorn Ospedale Dei Colli, Napoli
  - A.O.U. San Luigi Gonzaga, Orbassano
  - Istituto Oncologico Veneto, Padua
  - Azienda Ospedaliera Universitaria Di Parma, Parma
  - Policlinico San Matteo, Pavia
  - AUSL/IRCCS di Reggio Emilia, Reggio Emilia
  - IRCCS Regina Elena, Roma
  - Humanitas Cancer Center, IRCCS, Rozzano
  - Ospedale S. G. Moscati, Taranto
  - Azientda Sanitaria Universitaria Giuliano Isontina, Trieste